CLINICAL TRIAL: NCT01278342
Title: An Open-label, Two-step, Multicenter European Study to Evaluate the Efficacy and Safety of Sandostatin LAR at High Dose or in Combination Either With GH-receptor Antagonist or Dopamine-agonist in Acromegalic Patients Not Adequately Controlled by Conventional Regimen
Brief Title: Study to Evaluate the Efficacy and Safety of Sandostatin LAR at High Dose or in Combination Either With GH-receptor Antagonist or Dopamine-agonist in Acromegalic Patients
Acronym: HOSCAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995BIC03; 2005-005852-42 (Registry Identifier: EudraCT)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Results first posted 2011-02-17 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Acromegaly
Keywords: Sandostatin LAR; High Dose; GH-receptor antagonist; combination with dopamine-agonist; acromegalic patients; octreotide acetate; Somavert; Dostinex; pegvisomant; cabergoline; not adequately controlled; active acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide; pegvisomant; Cabergoline

ARMS (3):
- Sandostatin LAR high dose Alone (Active Comparator): All patients were treated with Sandostatin LAR 40 mg i.m. every 28 days for 3 months. Following biochemical assessment, patients with controlled GH and IGF-I after 3 months of Sandostatin LAR monotherapy continued to receive Sandostatin LAR 40 mg i.m. every 28 days for an additional 4 months.
  Interventions: Drug: Sandostatin LAR
- Sandostatin LAR high dose + Pegvisomat (Experimental): All patients were treated with Sandostatin LAR 40 mg i.m. every 28 days for 3 months. Following biochemical assessment, patients with uncontrolled GH and or IGF-I received Sandostatin LAR40 mg every 28 days in combination with weekly doses of pegvisomant 70 mg subcutaneously (s.c.) for a further 4 months
  Interventions: Drug: Sandostatin LAR; Drug: pegvisomant
- Sandostatin LAR high dose + Cabergoline (Experimental): All patients were treated with Sandostatin LAR 40 mg i.m. every 28 days for 3 months. Following biochemical assessment, patients with uncontrolled GH and or IGF-I received Sandostatin LAR 40 mg every 28 days in combination with weekly cabergoline for a further 4 months, with cabergoline doses as follows:
  1. st week: 0.25 mg twice a week (0.50 mg/week)
  2. nd week: 0.50 mg/week twice a week (1 mg/week)
  3. rd week: 0.50 mg four times a week (2 mg/week)
  4. th week: 0.50 mg daily (3.5 mg/week) Subsequent 3 months: 0.50 mg daily (3.5 mg/week)
  Interventions: Drug: Sandostatin LAR; Drug: cabergoline

INTERVENTIONS:
Drug: Sandostatin LAR — 40 mg intramuscular (i.m.) every 28 days for 3 months
  Other Names: octreotide acetate
Drug: pegvisomant — Weekly doses of pegvisomant 70 mg subcutaneously (s.c.) for 4 months given with Sandostatin LAR 40 mg intramuscular (i.m.) every 28 days for 4 months
  Other Names: Somavert; octreotide acaetate
  Arms: Sandostatin LAR high dose + Pegvisomat
Drug: cabergoline — Weekly cabergoline for 4 months, with weekly doses of Sandostatin LAR 40 mg intramuscular (i.m.) every 28 days for 4 months. Cabergoline doses as follows:
  1. st week: 0.25 mg twice a week (0.50 mg/week)
  2. nd week: 0.50 mg/week twice a week (1 mg/week)
  3. rd week: 0.50 mg four times a week (2 mg/week)
  4. th week: 0.50 mg daily (3.5 mg/week) Subsequent 3 months: 0.50 mg daily (3.5 mg/week)
  Other Names: Dostinex; octreotide acetate
  Arms: Sandostatin LAR high dose + Cabergoline

SUMMARY:
This study will assess the efficacy of 8 months treatment of Sandostatin® LAR® High Dose monotherapy or Sandostatin® LAR® High Dose in combination either with growth hormone antagonist or dopamine agonist to control biochemical parameters (GH and insulin-like growth factor I [IGF I]) of acromegalic patients not achieving biochemical normalization at conventional regimen.

ELIGIBILITY:
Inclusion Criteria:

• Patient with a biochemically documented active acromegaly, not adequately controlled by somatostatin-analogues at conventional regimen as follow : mean 1-hour GH > 2.5 ng/mL and elevated IGF-1 (adjusted for age and gender)

* Patient with reduction of either mean fasting GH at least 50% or IGF-1 at least 25% from any medical pretreatment level
* Patient currently receiving somatostatin-analogues at conventional regimen (maximum registered dose) for at least 6 months before inclusion

Exclusion Criteria:

* Newly diagnosed or previously medically untreated acromegalic patient
* Concomitant treatment with GH-receptor antagonist
* Concomitant treatment with dopamine-agonist
* Symptomatic cholelithiasis or choledocolithiasis
* Liver transaminases (ALT, AST) elevated, but > 3 times upper normal limit (according to local laboratory)
* Previous gamma-knife radiotherapy for treatment of acromegaly
* Compression of the optic chiasm causing visual field defect
* Any medical conditions contraindicated in the Summary of Product Characteristic (SPC) of all drugs

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- France (7):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
- Italy (7):
  - Novartis Investigative Site, Genova
  - Novarts Investigative Site, Naples
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Perugia
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Torino
- Poland (4):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
- Novartis Investigative Site, Porto, Portugal
- Novartis Investigative Site, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Sandostatin LAR High Dose + Pegvisomat: All patients were treated with Sandostatin LAR 40 mg i.m. every 28 days for 3 months. Following biochemical assessment, patients with uncontrolled GH and/or IGF-I, were randomized to receive Sandostatin LAR 40 mg every 28 days in combination with weekly doses of Pegvisomant 70 mg subcutaneously (s.c.) for a further 4 months.
- Sandostatin LAR High Dose + Cabergoline: All patients were treated with Sandostatin LAR 40 mg i.m. every 28 days for 3 months. Following biochemical assessment, patients with uncontrolled GH and/or IGF-I, were randomized to receive Sandostatin LAR 40 mg every 28 days in combination with weekly doses of Cabergoline for a further 4 months, with Cabergoline doses as follows:
  * 1st week: 0.25 mg twice a week (0.50 mg/week)
  * 2nd week: 0.50 mg/week twice a week (1 mg/week)
  * 3rd week: 0.50 mg four times a week (2 mg/week)
  * 4th week: 0.50 mg daily (3.5 mg/week) Subsequent 3 months: 0.50 mg daily (3.5 mg/week)
Period: Overall Study
Arm/Group | Sandostatin LAR High Dose Alone | Sandostatin LAR High Dose + Pegvisomat | Sandostatin LAR High Dose + Cabergoline
Started | 7 | 31 | 32
Completed | 3 | 30 | 32
Not Completed | 4 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Administrative problems | 2 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sandostatin LAR High Dose Alone | Sandostatin LAR High Dose + Pegvisomat | Sandostatin LAR High Dose + Cabergoline | Total
Number analyzed (Participants) | 7 | 31 | 32 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (7.71) | 44.6 (10.54) | 49.3 (10.50) | 48.1 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 17 | 18 | 38
  Male | 4 | 14 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Complete Response (CR) at 8 Months
Description: A patient was classified as a Complete Responder (CR) if both biochemical parameters were controlled at the end of 8 months of treatment:
  * Mean 1 hour GH < 2.5µg/L (according to Central Laboratory); and
  * IGF-I within the Central Laboratory Normal Range (for age and gender).
Time Frame: From Baseline to 8 months
Population: Intent-to-Treat population - all participants receiving at least one dose of Sandostatin LAR
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Sandostatin LAR High Dose Alone | Sandostatin LAR High Dose + Pegvisomat | Sandostatin LAR High Dose + Cabergoline
Number analyzed (Participants) | 7 | 31 | 32
percent | 25 [0.6 to 80.6] | 0 [0 to 11.2] | 9.4 [2.0 to 25.0]

2. Secondary Outcome: The Percentage of Participants With Complete Response (CR) At 3 Months
Description: A patient was classified as CR if both biochemical parameters were controlled at the end of 3 months of treatment:
  * Mean 1 hour GH < 2.5µg/L (according to Central Laboratory); and
  * IGF-I within the Central Laboratory Normal Range (for age and gender)
Time Frame: From Baseline to 3 months
Population: Intent-to-Treat population - all participants receiving at least one dose of Sandostatin LAR
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Sandostatin LAR High Dose Alone | Sandostatin LAR High Dose + Pegvisomat | Sandostatin LAR High Dose + Cabergoline
Number analyzed (Participants) | 7 | 31 | 32
percent | 60 [14.7 to 94.7] | 0 [0 to 11.2] | 0 [0 to 10.9]

3. Secondary Outcome: The Percentage of Participants With Partial Response (PR) at 8 Months
Description: Patients who met one of the following criteria at the end of 8 months of treatment were defined as Partial Responders, regardless of the treatment.
  * Mean 1 hour GH > 2.5 µg/L and < 5 µg/L and either a decrease in IGF-I of at least 50% compared to baseline or IGF-I within normal range.
  * Mean 1 hour GH < 2.5 µg/L and a decrease in IGF-I of at least 50% compared to baseline and IGF-I outside normal range.
Time Frame: From Baseline to 8 months
Population: Intent-to-Treat population - all participants receiving at least one dose of Sandostatin LAR
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Sandostatin LAR High Dose Alone | Sandostatin LAR High Dose + Pegvisomat | Sandostatin LAR High Dose + Cabergoline
Number analyzed (Participants) | 7 | 31 | 32
percent | 25 [0.6 to 80.6] | 22.6 [9.6 to 41.1] | 21.9 [9.3 to 40.0]

ADVERSE EVENTS:
Groups:
- Sandostatin LAR High Dose + Pegvisomant: All patients were treated with Sandostatin LAR 40 mg i.m. every 28 days for 3 months. Following biochemical assessment, patients with uncontrolled GH and/or IGF-I, were randomized to receive Sandostatin LAR 40 mg every 28 days in combination with weekly doses of Pegvisomant 70 mg subcutaneously (s.c.) for a further 4 months.
Arm/Group | Sandostatin LAR High Dose Alone | Sandostatin LAR High Dose + Pegvisomant | Sandostatin LAR High Dose + Cabergoline
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/32 | 2/31
Other Adverse Events (participants affected / at risk) | 4/7 | 15/32 | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sandostatin LAR High Dose Alone (N=7) | Sandostatin LAR High Dose + Pegvisomant (N=32) | Sandostatin LAR High Dose + Cabergoline (N=31)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sandostatin LAR High Dose Alone (N=7) | Sandostatin LAR High Dose + Pegvisomant (N=32) | Sandostatin LAR High Dose + Cabergoline (N=31)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 4 | 0
Blood insulin decreased (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Aphonia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 4
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.